CLINICAL TRIAL: NCT01679080
Title: The Effect of Treatment With Teriparatide and Zoledronic Acid in Patients With Osteogenesis Imperfecta
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Eli Lilly has withdrawn support to the study of teriparatide and placebo pens. The study was not able to continue as a randomized study without the supply of placebo pens.
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TreatOI
Record Dates: First submitted 2012-08-16; First posted 2012-09-05 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Osteogenesis Imperfecta
Keywords: Drug therapy; Adult
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Zoledronic Acid; Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zolendronic acid, 3 yr + placebo teriparatide, 2 yr (Experimental): yearly intravenous infusion of 5mg active zoledronic acid in 3 yr
  Interventions: Drug: Zoledronic acid
- teriparatide 2 yr; active zol in 3rd yr (Experimental): daily injection of one dose active teriparatide for two years, active zoledronic acid in year 3.
  Interventions: Drug: Zoledronic acid; Drug: Teriparatide
- No active treatment (Placebo Comparator): Observation in three years, no treatment
  Interventions: Other: No active treatment

INTERVENTIONS:
Drug: Zoledronic acid — antiresorptive and calcium and vitamin D
  Other Names: zolendronate; Aclasta
  Arms: Zolendronic acid, 3 yr + placebo teriparatide, 2 yr; teriparatide 2 yr; active zol in 3rd yr
Drug: Teriparatide — anabolic and calcium and vitamin D
  Other Names: PTH; Forsteo
  Arms: teriparatide 2 yr; active zol in 3rd yr
Other: No active treatment — Calcium and vitamin D
  Arms: No active treatment

SUMMARY:
Osteogenesis imperfecta (OI) is an inherited disease of the connective tissue. Symptoms are fractures, growth retardation, blue sclera, bad teeth, impaired hearing a.o. The aim of the present study is to investigate the effect of treatment of adult OI patients with bisphosphonate (zoledronic acid), parathyroid hormone (PTH) or placebo on bone mass, fracture risk and quality of life.

The investigators will therefore conduct a double blind, placebo controlled trial, taking genotype and previous antiresorptive therapy into account.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of osteogenesis imperfecta
* BMD<-1.0 or

Exclusion Criteria:

* creatinine clearance <30mL/min
* treatment with glucocorticoids > 5mg daily during the last 3 months
* metabolic bone disease or vitamin d deficiency
* liver or kidney disease
* contradictions to zoledronic acid or teriparatide
* increased baseline risk of osteosarcoma

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-11; Primary Completion 2020-07-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) | Three years
  Dual-energy X-ray absorptiometry scans are performed at the lumbar spine, hip and whole body twice yearly. The value of the lumbar BMD is the primary outcome.

SECONDARY OUTCOMES:
Fracture risk | Three years
  Participants are asked to report fractures throughout the study. Medical examination yearly with a focus on possible new fractures. Columnar x-ray before and after the study investigate new fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Langdahl, MD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Osteoporosis clinic; department of endocrinology and metabolism, Aarhus, Aarhus C
  - Department of endocrinology, Hvidovre
  - Department of Endocrinology M, Odense